CLINICAL TRIAL: NCT03253250
Title: A Prospective, Randomized, Multicenter, Open-label, Exploratory Study of Utilizing of Peginterferon Alfa-2a on the Relapse Rate of the Subjects With Hepatocellular Carcinoma Who Have Been Treated by Resection
Brief Title: The Investigation of Peginterferon Alfa-2a on the RFS of the Subjects With HCC Who Have Been Treated by Resection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jiming Zhang, Deputy director of department, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEG-HCC
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Chronic Hepatitis b; Hepatic Carcinoma
MeSH Terms: conditions — Hepatitis B, Chronic; Carcinoma, Hepatocellular | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): The subjects will be treated by NAs (ETV, 0.5mg，qd；TDF，300mg，qd；ADV，10mg，qd）for 96 weeks
  Interventions: Drug: ETV；TDF；ADV
- Group B (Experimental): The subjects will be treated by peginterferon alfa-2a （135μg/week）combination with NAs(ETV\TDF\ADV) for 96 weeks.
  Interventions: Drug: ETV；TDF；ADV; Drug: Peginterferon Alfa-2a

INTERVENTIONS:
Drug: ETV；TDF；ADV — NAs
  Other Names: entecavir;tenofovir disoproxil fumarate;adefovir
Drug: Peginterferon Alfa-2a — peginterferon
  Other Names: pegasys
  Arms: Group B

SUMMARY:
The current study is a prospective, randomized, open, multi-center investigation. The aim of current study is to investigate whether the Recurrence-free Survival Rate (RFS）of the hepatitis B related -hepatocellular carcinoma subjects who have been treated by resection can be improved by peginterferon alfa-2a

DETAILED DESCRIPTION:
The subjects who have been treated by resection due to hepatocellular carcinoma (HCC) will be randomized into 2 groups: the subjects in group A will be treated by Nucleotide analogues (NAs)( ETV, 0.5mg，qd；tenofovir disoproxil fumarate(TDF)，300mg，qd；ADV，10mg，qd）for 96 weeks; the subjects in group B will be treated by peginterferon alfa-2a （135μg/week）combination with NAs (ETV\TDF\ADV)for 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients with age ≥18 and ≤70 years;
2. Expected survival time >3 months;
3. There should be evidences that chronic hepatitis B or hepatitis have been positive, hepatitis B virus (HBV) DNA detectable or undetectable, Alanine aminotransferase(ALT)<upper limit of normal (ULN) or ≥ULN；
4. The patients have been treated by resection due to HCC;
5. The characteristic of tumor should be:Barcelona Clinic Liver Cancer(BCLC): 0,A,B
6. Child-Pugh scores:A
7. Agree to participate in the study and sign the patient informed consent form.

Exclusion Criteria:

1. Patients that have been treated by live transplantation、chemoembolization、radiotherapy、chemotherapy、molecular targeted therapy and biotherapy before the resection;
2. Patients that are treated by hepatotoxicity drugs 、immunosuppressant or adjuvant chemotherapy after the resection;
3. Patients who be treated by transcatheter arterial chemoembolization(TACE) after resection;
4. BCLC(Barcelona Clinic Liver Cancer):C、D before the resection;
5. History or other evidence of malignant tumor: except by basal cell carcinoma or squamous cell carcinoma which are cured 、carcinoma in situs of cervix
6. Allergic history to interferon;
7. Co-infection with active hepatitis A, hepatitis C, hepatitis D and/or human immunodeficiency virus (HIV);
8. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
9. absolute neutrophil count(ANC)<1.5x 10^9/L or platelet count(PLT)<70x 10^9/L
10. Creatinine over upper limit of normal;
11. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as major depression or psychosis that treated with antidepressant medication or a major tranquilizer at therapeutic doses respectively at any time prior to 3 months or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
12. History of severe cardiac disease (e.g., New York Heart Association Functional Class III or IV, myocardial infarction within 6 months, ventricular tachyarrhythmias requiring ongoing treatment, unstable angina or other significant cardiovascular diseases);
13. History of thyroid disease poorly controlled on prescribed medications;
14. Evidence of severe retinopathy or clinically relevant ophthalmologic disorder;
15. History of other severe disease or evidence of other severe disease or any other illness or conditions that the investigator believe that patients are not suitable to join in the study;
16. Evidence of postoperative complications: infectious、bleeding, etc,. at baseline; or evidence of recurrence or metastasis at baseline;
17. Child-Pugh scores :B、C
18. Patients included in another trial or having been given investigational drugs within 12 weeks prior to screening;
19. Other disease should exclusive considered by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free Survival Rate (RFS） | 2 years
  Number of subjects without Recurrence in the total subjects

SECONDARY OUTCOMES:
Recurrence-free Survival Rate (RFS） | 1 year
  Number of subjects without Recurrence in the total subjects
Overall Survival Rate (OS） | 2 years
  Number of subjects with survival in the total subjects
Overall Survival Rate (OS） | 1 year
  Number of subjects with survival in the total subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lunxiu Qin, Principal Investigator — Huashan Hospital; Jimimg Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China

REFERENCES:
- [Background] Sun HC, Tang ZY, Wang L, Qin LX, Ma ZC, Ye QH, Zhang BH, Qian YB, Wu ZQ, Fan J, Zhou XD, Zhou J, Qiu SJ, Shen YF. Postoperative interferon alpha treatment postponed recurrence and improved overall survival in patients after curative resection of HBV-related hepatocellular carcinoma: a randomized clinical trial. J Cancer Res Clin Oncol. 2006 Jul;132(7):458-65. doi: 10.1007/s00432-006-0091-y. Epub 2006 Mar 24. PMID 16557381
- [Background] Sohn W, Paik YH, Kim JM, Kwon CH, Joh JW, Cho JY, Gwak GY, Choi MS, Lee JH, Koh KC, Paik SW, Yoo BC. HBV DNA and HBsAg levels as risk predictors of early and late recurrence after curative resection of HBV-related hepatocellular carcinoma. Ann Surg Oncol. 2014 Jul;21(7):2429-35. doi: 10.1245/s10434-014-3621-x. Epub 2014 Mar 12. PMID 24619495
- [Background] Micco L, Peppa D, Loggi E, Schurich A, Jefferson L, Cursaro C, Panno AM, Bernardi M, Brander C, Bihl F, Andreone P, Maini MK. Differential boosting of innate and adaptive antiviral responses during pegylated-interferon-alpha therapy of chronic hepatitis B. J Hepatol. 2013 Feb;58(2):225-33. doi: 10.1016/j.jhep.2012.09.029. Epub 2012 Oct 6. PMID 23046671